CLINICAL TRIAL: NCT02634723
Title: Retrospective Chart Review to Evaluate Safety and Tolerability of ADVATE Among Previously Untreated Patients in China With Moderate to Severe Hemophilia A
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 061501
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Previously Untreated Patients (PUPs): PUPs in China with Moderate to Severe Hemophilia A
  Interventions: Biological: Octocog alfa (recombinant human coagulation factor VIII)

INTERVENTIONS:
Biological: Octocog alfa (recombinant human coagulation factor VIII)
  Other Names: ADVATE; Recombinant antihemophilic factor; plasma/albumin-free method (rAHF-PFM

SUMMARY:
The purpose of this post-marketing safety study is to evaluate the safety, immunogenicity, and effectiveness of ADVATE in previously untreated patients (PUPs) in China with moderate to severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated patient (PUP) in China with moderate to severe hemophilia A.
2. Investigator prescribed ADVATE as the predominant therapeutic agent for the management of hemophilia A
3. Informed consent form from patient and/or legal representative will need to be signed per local regulation

Exclusion Criteria:

1. Presence of an inherited or acquired hemostatic defect other than hemophilia A, and any other clinically significant chronic disease
2. Participants who participated in another investigational FVIII drug study, or had participated in any clinical study involving an investigational FVIII drug during the course of the observation period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously untreated patients (PUPs) in China with moderate to severe hemophilia A.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Number of high titer, low titer and transient Factor VIII (FVIII) inhibitors developed | Throughout the study period of 6 months
Number and type of other serious and non-serious adverse events (AEs) | Throughout the study period of 6 months
  Other AEs refers to AEs other than Factor VIII (FVIII) inhibitors

SECONDARY OUTCOMES:
Number and type of bleeding episodes treated with ADVATE | Throughout the study period of 6 months
Number of bleeding episodes treated with 1, 2, 3, ≥ 4 infusions of ADVATE | Throughout the study period of 6 months
Annualized bleeding rate (ABR) of participants treated prophylactically and on-demand with ADVATE | Throughout the study period of 6 months
Annualized joint bleeding rate (AJBR) of participants treated prophylactically and on-demand with ADVATE | Throughout the study period of 6 months
Total number of exposure days (EDs) to ADVATE | Throughout the study period of 6 months
Total units of ADVATE administered | Throughout the study period of 6 months
Total number of exposure days (EDs) to all Factor VIII (FVIII) products | Throughout the study period of 6 months
Total units of all Factor VIII (FVIII) products administered | Throughout the study period of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- China (6):
  - Institute of Hematology and Oncology, Harbin The First Hospital, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Nanjing Children's Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Shandong Blood Center, Jinan, Shandong
  - Zhejiang Provincial Hospital of TCM/The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc24db2bf003ab45811